CLINICAL TRIAL: NCT03155191
Title: A Multicenter Phase I/II Study for Relapsed or Refractory CD19+ B-acute Lymphoblastic Leukemia
Brief Title: Study of TBI-1501 for Relapsed or Refractory Acute Lymphoblastic Leukemia
Acronym: TBI-1501
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501-01
Record Dates: First submitted 2017-04-14; First posted 2017-05-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Lymphoblastic Leukemia, Acute Adult
Keywords: Acute lymphoblastic leukemia; Leukemia; Lymphoblastic; TBI-1501; Anti-CD19 CAR Expressing T cells Therapy; CD19 CAR Gene-Transduced Lymphocyte; Adoptive Immunotherapy; Genetically Engineered Lymphocyte Therapy; Retroviral Vector; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases; Chimeric antigen receptor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Peripheral blood will be collected from a subject after obtaining a written informed consent. Peripheral blood mononuclear cells (PBMCs) and plasma are obtained from the blood, and T cells contained in the PBMCs are transduced with anti-CD19 CAR gene by using retroviral vector.
  Cyclophosphamide will be administered after obtaining a written informed consent and completing registration.
  CD19-CAR-T will be administered in the split dose. Phase 2 recommended dose will be applied for phase 1 portion. The investigator assesses efficacy of CD19-CAR-T in accordance with study-specific criteria, at 8 week after the infusion of CD19-CAR-T (or at the time of termination). The investigator also assesses the safety during the follow-up period. Long-term follow-up study is conducted at frequency of once a year for 15 years after the infusion of CD19-CAR-T in reference to guidelines of FDA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Level -1 to 2 (Experimental): 0.3 to 3 x 10^6 autologous CD19-CAR-T cells/kg per patient will be administered intravenously after a conditioning chemotherapy with cyclophosphamide.
  cohort -1: 3×10^5 cells/kg cohort 1: 1×10^6 cells/kg cohort 2: 3×10^6 cells/kg.
  Interventions: Biological: TBI-1501

INTERVENTIONS:
Biological: TBI-1501 — Phase-I portion:
  Cyclophosphamide is administered for conditioning medication of TBI1501, that is CD19-CAR-T cells, (cohort -1: 3×10^5 cells/kg, cohort 1: 1×10^6 cells/kg, cohort 2: 3×10^6 cells/kg).
  Phase-II portion:
  Recommended dose of Phase-II part will be administered. Cyclophosphamide will be administered as conditioning. The end of study will be Week 52 after administration of TBI-1501.

SUMMARY:
Evaluate the safety (P-I), pharmacokinetics and anti-tumor effect of immunotherapy of autologous T cells genetically modified to express anti-CD19 chimeric antigen receptor (CAR) (TBI-1501) for relapsed or refractory CD19+ B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Enroll patients after confirming eligibility. Following enrollment, peripheral blood mononuclear cells and blood plasma will be obtained from each subject by apheresis to start the manufacturing of TBI-1501.

Before TBI-1501 administration, it is necessary to pass the quality tests. Subject will be hospitalized from Day -3 to Day 28, and administered Cyclophosphamide (1,000 mg/m2/day×2 days) on Day -3 and Day -2.

ELIGIBILITY:
Inclusion Criteria:

1. In phase-1 study, patients must be ≥ 18 years of age. In phase-2 study, patients must be ≥ 16 years of age.
2. Patients with relapse or refractory CD19+ acute B-cell lymphoblastic leukemia
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
4. Patients must have adequate key organ function (bone marrow, heart, lung, liver, renal, etc), as defined below

   * Total bilirubin level ≤1.5xULN (Upper limit of normal)
   * AST(GOT)/ALT(GPT) level ≤5.0xULN
   * Serum creatinine ≤2.0mg/dL
   * SpO2 ≧ 92%
   * LVEF ≥50%
5. Patients must be able to understand and willing to sign a written informed consent document (for patients <20 years of age their legal guardian must give informed consent).

Exclusion Criteria:

1. White blood cell counts ≧ 50,000/uL
2. Received expected antitumor therapy (chemotherapy or radiation therapy, etc) within 2 weeks.
3. Received HSCT within 12 weeks before enrollment.
4. Under treatment for GVHD.
5. lymphocytes except for blasts ≦ 500/uL
6. Presence of active CNS-3
7. Concurrent use of systemic steroids or immunosuppressive agents (except for replacement therapy and local administration. e.g. inhalation, application and so on).
8. HBs Ag positive ,or either HBc Ab positive or HBs positive with HBV-DNA > 1.3LogIU/ml
9. Presence of active hepatitis C infection
10. HIV Ab or anti-HTLV-1 Ab positive
11. History of allergy about component of investigational product or animal(cattle and/or mouse)-derived additives
12. Hypersensitivity to antibiotics.
13. Presence of symptomatic cardiac arrhythmias or serious heart disease.
14. Presence of another malignant tumor.
15. Psychiatric disorder, alcohol addiction or drug addiction that affects the ability of informed consent.
16. Active or serious infection.
17. Both men and women who have generative functions, and who cannot agree with using contraceptive devices from the day of the consent to the end of study.
18. Pregnant or lactating women.
19. Any other patients judged by the investigators to be inappropriate for the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2035-03-31 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase-I portion: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | One year
  Adverse event (frequency, seriousness, duration, causality, severity, classification), mortality, severe adverse event, discontinuation due to adverse event.
Phase-II portion: Anti-tumor effect (CR+CRi rate) | 56 days
  Complete Remission (CR)+Complete Remission with Incomplete Blood Count Recovery (CRi) , as determined by assessments of peripheral blood and bone marrow.

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Akita University Hospital, Akita, Akita
  - University Of Fukui Hospital, Yoshida, Fukui
  - Kyushu University Hospital, Higashiku, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Jichi Medical University hospital, Shimotsuke-shi, Tochigi
  - Cancer Institute Hospital Of JFCR, Kōto, Tokyo
  - The Institute of Medical Science, The University of Tokyo, Minato-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No